CLINICAL TRIAL: NCT00114517
Title: Biologic Response of Menopausal Women to 17B-Estradiol
Brief Title: ELITE: Early Versus Late Intervention Trial With Estradiol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Howard N. Hodis, M.D., Harry J. Bauer and Dorothy Bauer Rawlins Professor of Cardiology, Professor of Medicine, Population and Public Health Sciences, and Molecular Pharmacology and Toxicology, Director, Atherosclerosis Research Unit, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AG0025; R01AG024154 (NIH)
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; CAD; cardiac computed tomography; cardiovascular disease; carotid artery intima-media thickness; cognitive function; computed tomography; coronary artery calcium; coronary artery disease; coronary artery lesions; CVD; estrogen; estrogen therapy; hormone therapy; postmenopausal; subclinical vascular disease; timing hypothesis; ultrasonography; menopausal hormone replacement therapy; menopause; prevention; intervention
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease | interventions — Estradiol; Estrogens; Estrogen Replacement Therapy; Hormone Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 17B-estradiol (Active Comparator): Oral 17B-estradiol 1 mg daily
  Interventions: Drug: 17B-estradiol
- Placebo (Placebo Comparator): Matching oral 17B-estradiol placebo daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 17B-estradiol — Oral 17B-estradiol 1 mg daily
  Other Names: Estrace; Estrogen; Estrogen replacement therapy; Hormone replacement therapy; Hormone therapy; Menopausal hormone replacement therapy
  Arms: 17B-estradiol
Other: Placebo — Matching oral 17B-estradiol placebo daily
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of oral 17B-estradiol (estrogen) on the progression of early (subclinical) atherosclerosis and cognitive decline in healthy postmenopausal women.

DETAILED DESCRIPTION:
The primary hypothesis to be tested is that 17B-estradiol (estrogen) will reduce the progression of early atherosclerosis if initiated soon after menopause when the vascular endothelium (lining of blood vessels) is relatively healthy versus later when the endothelium has lost its responsiveness to estrogen. Ultrasonography will be used to measure the rate of change in the thickness of the carotid artery and cardiac computed tomography (CT) will be used to measure coronary artery calcium and coronary artery lesions. The second hypothesis to be tested is that 17B-estradiol (estrogen) will reduce the progression of cognitive decline if initiated soon after menopause when healthy brain tissue remains responsive to estrogen versus later when brain tissue has lost its responsiveness to estrogen.

A total of 643 (actual; 504 initially proposed) postmenopausal women were randomized according to their number of years since menopause, less than 6 years or 10 years or more, to receive either oral 17B-estradiol 1 mg daily or matching placebo. Women with a uterus will also use vaginal progesterone gel 4% (or placebo gel) the last ten days of each month. The vaginal progesterone will be distributed in a double-blinded fashion along with the randomized treatment so that only women exposed to active treatment will receive active progesterone. As initially proposed, participants will undergo ultrasonography at baseline and every 6 months throughout the 2 to 5 years (average 3 years) of randomized treatment. Participants will also undergo cognitive testing at baseline and after 3 years of randomized treatment. The trial has been extended for an additional 2 to 2.5 years of randomized treatment (overall average randomized treatment of 5 years and range of 2 to 8.5 years). Ultrasonography will continue to be collected every 6 months and upon completion of randomized treatment, participants will undergo cardiac CT for coronary artery calcium and coronary artery lesion measurements. Participants will also undergo a third cognitive testing at the completion of randomized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women with a serum estradiol level 25 pg/ml or less
* No period for 6 months or more
* Postmenopausal less than 6 years, OR 10 years or longer

Exclusion Criteria:

* Clinical signs, symptoms, or personal history of cardiovascular disease
* Women who have had a hysterectomy only and no oophorectomy (since time from menopause cannot be determined)
* Diabetes mellitus or fasting serum glucose 140 mg/dL or greater
* Uncontrolled hypertension (diastolic blood pressure 110 mmHg or greater)
* Thyroid disease (untreated)
* Serum creatinine greater than 2.0 mg/dL
* Plasma triglyceride levels greater than 500 mg/dL
* Life threatening disease with prognosis less than 5 years
* Cirrhosis or liver disease
* History of deep vein thrombosis or pulmonary embolism
* History of breast cancer
* Current hormone replacement therapy (HRT)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2004-07; Primary Completion 2013-02-12 (Actual); Study Completion 2013-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, M.D., Principal Investigator — Atherosclerosis Research Unit, University of Southern California
Locations (1):
- Atherosclerosis Research Unit, University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Background] Hodis HN, Mack WJ, Shoupe D, Azen SP, Stanczyk FZ, Hwang-Levine J, Budoff MJ, Henderson VW. Methods and baseline cardiovascular data from the Early versus Late Intervention Trial with Estradiol testing the menopausal hormone timing hypothesis. Menopause. 2015 Apr;22(4):391-401. doi: 10.1097/GME.0000000000000343. PMID 25380275
- [Result] Hodis HN, Mack WJ, Henderson VW, Shoupe D, Budoff MJ, Hwang-Levine J, Li Y, Feng M, Dustin L, Kono N, Stanczyk FZ, Selzer RH, Azen SP; ELITE Research Group. Vascular Effects of Early versus Late Postmenopausal Treatment with Estradiol. N Engl J Med. 2016 Mar 31;374(13):1221-31. doi: 10.1056/NEJMoa1505241. PMID 27028912
- [Result] Henderson VW, St John JA, Hodis HN, McCleary CA, Stanczyk FZ, Shoupe D, Kono N, Dustin L, Allayee H, Mack WJ. Cognitive effects of estradiol after menopause: A randomized trial of the timing hypothesis. Neurology. 2016 Aug 16;87(7):699-708. doi: 10.1212/WNL.0000000000002980. Epub 2016 Jul 15. PMID 27421538
- [Derived] Chen IJ, Stanczyk FZ, Sriprasert I, Karim R, Shoupe D, Kono N, Hodis HN, Mack WJ. Sex steroid hormones and subclinical atherosclerosis progression in postmenopausal women. Eur J Endocrinol. 2025 Mar 3;192(3):248-256. doi: 10.1093/ejendo/lvaf032. PMID 39980346
- [Derived] Lin F, Pa J, Karim R, Hodis HN, Han SD, Henderson VW, St John JA, Mack WJ. Subclinical carotid artery atherosclerosis and cognitive function in older adults. Alzheimers Res Ther. 2022 May 7;14(1):63. doi: 10.1186/s13195-022-00997-7. PMID 35526057
- [Derived] Sriprasert I, Mert M, Mack WJ, Hodis HN, Shoupe D. Use of oral estradiol plus vaginal progesterone in healthy postmenopausal women. Maturitas. 2021 Dec;154:13-19. doi: 10.1016/j.maturitas.2021.09.002. Epub 2021 Sep 5. PMID 34736575
- [Derived] Sriprasert I, Kono N, Karim R, Hodis HN, Stanczyk FZ, Shoupe D, Mack WJ. Factors Associated With Serum Estradiol Levels Among Postmenopausal Women Using Hormone Therapy. Obstet Gynecol. 2020 Oct;136(4):675-684. doi: 10.1097/AOG.0000000000004006. PMID 32925623
- [Derived] Sriprasert I, Mack WJ, Hodis HN, Allayee H, Brinton RD, Karim R. Effect of ApoE4 Genotype on the Association Between Metabolic Phenotype and Subclinical Atherosclerosis in Postmenopausal Women. Am J Cardiol. 2019 Oct 1;124(7):1031-1037. doi: 10.1016/j.amjcard.2019.06.022. Epub 2019 Jul 15. PMID 31362877
- [Derived] Sriprasert I, Hodis HN, Karim R, Stanczyk FZ, Shoupe D, Henderson VW, Mack WJ. Differential Effect of Plasma Estradiol on Subclinical Atherosclerosis Progression in Early vs Late Postmenopause. J Clin Endocrinol Metab. 2019 Feb 1;104(2):293-300. doi: 10.1210/jc.2018-01600. PMID 30272234
- [Derived] Karim R, Stanczyk FZ, Brinton RD, Rettberg J, Hodis HN, Mack WJ. Association of endogenous sex hormones with adipokines and ghrelin in postmenopausal women. J Clin Endocrinol Metab. 2015 Feb;100(2):508-15. doi: 10.1210/jc.2014-2834. Epub 2014 Nov 18. PMID 25405497
- [Derived] Henderson VW. Aging, estrogens, and episodic memory in women. Cogn Behav Neurol. 2009 Dec;22(4):205-14. doi: 10.1097/WNN.0b013e3181a74ce7. PMID 19996872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population through media campaigns.
Pre-assignment Details: 2166 individuals were screened by telephone, 1,271 were ineligible. 895 individuals were screened in research clinic, 252 were excluded (133 did not meet inclusion criteria; 119 declined to participate). 643 individuals were randomized.
Groups:
- Early Postmenopause 17B-estradiol: Early postmenopause, <6 years-since-menopause, Oral 17B-estradiol 1 mg daily
- Early Postmenopause Placebo: Early postmenopause, <6 years-since-menopause, Matching oral 17B-estradiol placebo daily
- Late Postmenopause 17B-estradiol: Late postmenopause, >10 years-since-menopause, Oral 17B-estradiol 1 mg daily
- Late Postmenopause Placebo: Late postmenopause, >10 years-since-menopause, Matching oral 17B-estradiol placebo daily
Period: Overall Study
Arm/Group | Early Postmenopause 17B-estradiol | Early Postmenopause Placebo | Late Postmenopause 17B-estradiol | Late Postmenopause Placebo
Started | 137 | 134 | 186 | 186
Completed | 125 | 123 | 172 | 176
Not Completed | 12 | 11 | 14 | 10
Not completed — Adverse Event | 6 | 1 | 6 | 3
Not completed — Lost to Follow-up | 2 | 2 | 2 | 1
Not completed — Too busy | 3 | 1 | 1 | 2
Not completed — Moved from area | 0 | 3 | 2 | 1
Not completed — Did not want estradiol | 1 | 1 | 0 | 0
Not completed — Armed-services duty | 0 | 1 | 0 | 1
Not completed — Competing family issue | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Lost interest | 0 | 0 | 1 | 0
Not completed — Weight increase | 0 | 0 | 1 | 0
Not completed — Concern about blood clots | 0 | 0 | 1 | 0
Not completed — Breast cancer diagnosis on baseline mammogram | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Postmenopause 17B-estradiol | Early Postmenopause Placebo | Late Postmenopause 17B-estradiol | Late Postmenopause Placebo | Total
Number analyzed (Participants) | 125 | 123 | 172 | 176 | 596
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.4 [53.2 to 57.9] | 55.4 [52.5 to 57.8] | 64.3 [60.5 to 68.6] | 63.0 [59.9 to 67.0] | 60.0 [55.5 to 64.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 123 | 172 | 176 | 596
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-hispanic | 88 | 73 | 127 | 127 | 415
  Black, non-hispanic | 7 | 14 | 17 | 14 | 52
  Hispanic | 16 | 20 | 20 | 23 | 79
  Asian | 14 | 16 | 8 | 12 | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression of Subclinical Atherosclerosis
Description: Rate of change in distal common carotid artery (CCA) far wall intima-media thickness (mm per year) in computer image processed B-mode ultrasonograms that were obtained at two baseline examinations (averaged to obtain the baseline CIMT value) and every 6 months during trial follow-up.
Time Frame: Baseline x 2 and then every 6 months up to 6.7 years
Population: Early postmenopause group (<6 years-since-menopause) at baseline and late postmenopause group (>10 years-since-menopause) at baseline.
Measure: Mean (95% Confidence Interval); unit: mm per year
Arm/Group | 17B-estradiol | Placebo
Number analyzed (Participants) | 297 | 299
mm per year
  Early postmenopause group: number analyzed (Participants) | 125 | 123
  Early postmenopause group | 0.0044 [0.0026 to 0.0061] | 0.0078 [0.0060 to 0.0096]
  Late postmenopause group: number analyzed (Participants) | 172 | 176
  Late postmenopause group | 0.0100 [0.0085 to 0.0115] | 0.0088 [0.0073 to 0.0103]

2. Secondary Outcome: Change in Neurocognitive Function (Global Cognition)
Description: All neuropsychological test scores at baseline and follow-up assessments were standardized ([raw score - mean score]/standard deviation) using the baseline means and standard deviations from the entire ELITE sample. Each of three cognitive composite scores was calculated at baseline and follow-up assessments as the weighted average of the individual donor standardized test scores, weighted by the inverse correlation among tests.The change from baseline (endpoint minus baseline cognitive outcome) was computed for each of the cognitive scores (verbal memory, global cognition, and executive functions). Since the outcome is not a single test but a weighted average of multiple tests, the range is not standard and not reported. Higher scores mean better outcomes.
Time Frame: Baseline and at 2.5 years and 5 years
Population: Sample size represents the number of participants with analyzable data collected at baseline, 2.5 years, and 5.0 years. Early postmenopause group (<6 years-since-menopause) at baseline and late postmenopause group (>10 years-since-menopause) at baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 17B-estradiol | Placebo
Number analyzed (Participants) | 284 | 283
units on a scale
  Early postmenopause group: number analyzed (Participants) | 121 | 113
  Early postmenopause group | 0.42 [0.11 to 0.73] | 0.40 [-0.07 to 0.72]
  Late postmenopause group: number analyzed (Participants) | 163 | 170
  Late postmenopause group | 0.29 [0.14 to 0.44] | 0.36 [0.20 to 0.53]

3. Secondary Outcome: Coronary Artery Calcium
Description: Number of participants with coronary artery calcium measured by cardiac computed tomography
Time Frame: End of randomized treatment, up to 6.7 years
Population: CAC data was obtained in 380 participants. Participants who were not taking the study products at the last follow-up visit, who had adherence to the study regimen that was lower than 80%, or who had a CAC scan more than 6 months after the final study visit were not included in the analysis. Early postmenopause group (<6 years-since-menopause) at baseline and late postmenopause group (>10 years-since-menopause) at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | 17B-estradiol | Placebo
Number analyzed (Participants) | 188 | 192
Participants
  Early postmenopause group: number analyzed (Participants) | 87 | 79
  Early postmenopause group | 34 | 24
  Late postmenopause group: number analyzed (Participants) | 101 | 113
  Late postmenopause group | 57 | 65

ADVERSE EVENTS:
Description: Adverse events collected per intervention
Arm/Group | 17B-estradiol | Placebo
All-Cause Mortality (participants affected / at risk) | 1/323 | 1/320
Serious Adverse Events (participants affected / at risk) | 43/323 | 45/320
Other Adverse Events (participants affected / at risk) | 216/323 | 226/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 17B-estradiol (N=323) | Placebo (N=320)
aplastic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
unstable angina (Cardiac disorders) | 2 (2) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
veritgo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
ischemic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
illeitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
death (General disorders) | 1 (1) | 1 (1)
non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
cellulitis (Infections and infestations) | 0 (0) | 2 (2)
lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 1 (1)
cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
polycythemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
amnesia (Nervous system disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 1 (1)
transient ischemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Suicide ideation (Psychiatric disorders) | 0 (0) | 1 (1)
psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
ulcerative colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 17B-estradiol (N=323) | Placebo (N=320)
chest discomfort (General disorders) | 23 (23) | 22 (22)
non-cardiac chest pain (General disorders) | 18 (18) | 12 (12)
drug hypersensitivity (Immune system disorders) | 26 (26) | 25 (25)
bronchitis (Infections and infestations) | 19 (19) | 22 (22)
influenza (Infections and infestations) | 44 (44) | 52 (52)
sinusitis (Infections and infestations) | 24 (24) | 24 (24)
urinary tract infection (Infections and infestations) | 63 (63) | 64 (64)
contusion (Injury, poisoning and procedural complications) | 17 (17) | 12 (12)
fall (Injury, poisoning and procedural complications) | 37 (37) | 36 (36)
road traffic accident (Injury, poisoning and procedural complications) | 19 (19) | 13 (13)
arthralgia (Musculoskeletal and connective tissue disorders) | 47 (47) | 53 (53)
back pain (Musculoskeletal and connective tissue disorders) | 35 (35) | 32 (32)
pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 18 (18)
depression (Psychiatric disorders) | 17 (17) | 20 (20)
cervical dysplasia (Reproductive system and breast disorders) | 48 (48) | 42 (42)
vaginal discharge (Reproductive system and breast disorders) | 17 (17) | 8 (8)
vulvovaginal pruritis (Reproductive system and breast disorders) | 19 (19) | 11 (11)
cough (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 19 (19)
rash (Skin and subcutaneous tissue disorders) | 16 (16) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No